CLINICAL TRIAL: NCT05921981
Title: Comparison of the Effectiveness of White Noise and Multisensory Stimulation in Retinopathy Examination
Brief Title: Multisensory Stimulation Versus White Noise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Halil Ibrahim Tasdemir, Assistant Professor, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MAKU23-368
Record Dates: First submitted 2023-06-19; First posted 2023-06-27 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Retinopathy; Premature Retinopathy
Keywords: preterm infants; Multisensorial stimulation; White Noise
MeSH Terms: conditions — Retinal Diseases; Retinopathy of Prematurity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multisensorial Stimulation Group (Experimental): The group to which multi-sensory stimulation will be applied during the retinopathy examination.
  Interventions: Behavioral: Multisensorial Stimulation
- White Noise Group (Active Comparator): The group to which White Noise will be applied during the retinopathy examination.
  Interventions: Behavioral: White Noise
- Control Group (No Intervention): The group that will receive routine care during the retinopathy examination

INTERVENTIONS:
Behavioral: Multisensorial Stimulation — Multisensory stimulation in newborns involves the deliberate and simultaneous activation of multiple sensory modalities to provide sensory experiences that promote development and enhance learning. Newborns are naturally inclined to explore and make sense of their environment through their senses, including touch, sight, sound, taste, and smell.
  Arms: Multisensorial Stimulation Group
Behavioral: White Noise — White Noise
  Arms: White Noise Group

SUMMARY:
This study aimed to compare the effectiveness of two interventions, white noise, and multisensory stimulation, during retinopathy examinations on premature infants. Retinopathy is a common eye disorder among premature infants, which can cause visual impairments if not addressed. The research used a randomized controlled experimental design, with premature infants randomly assigned to either the white noise or multisensory stimulation group or control group. Physiological responses, behavioral indicators, and the pain of the retinopathy examination were measured. Trained healthcare professionals conducted the investigations in a controlled environment, and statistical analyses were employed to compare the outcomes between the three groups. The findings of this study have the potential to inform the development of more effective and well-tolerated examination protocols for premature infants, leading to improved visual outcomes and overall well-being for this vulnerable population.

DETAILED DESCRIPTION:
This study aimed to compare the effectiveness of white noise and multisensory stimulation in retinopathy examination on premature infants. Retinopathy is a common eye disorder among premature infants that can lead to long-term visual impairments if left untreated. Therefore, finding effective interventions for retinopathy examinations is crucial for improving the overall visual health of these infants.

A randomized controlled experimental design was employed, with premature infants as the study participants. The infants were randomly assigned to three groups: the control group, the white noise group, and the multisensory stimulation group. The white noise group received auditory stimulation through the presentation of white noise, while the multisensory stimulation group received additional visual and tactile stimuli during the retinopathy examination.

Several outcome measures were used to evaluate the effectiveness of the interventions. These measures included physiological responses (e.g., heart rate, blood pressure), behavioral indicators (e.g., eye movement, crying), and overall examination success rate. The examination success rate was defined as the ability to complete the retinopathy examination without disturbances caused by infant distress or movement.

The study employed trained healthcare professionals who performed retinopathy examinations using standardized procedures. Data collection was conducted in a controlled environment to ensure consistency across three groups. Statistical analyses, such as ANOVA and chi-square tests, were employed to compare the outcomes between the three groups.

The findings of this study have the potential to contribute to the development of effective and well-tolerated retinopathy examination protocols for premature infants. By comparing the effects of white noise and multisensory stimulation, the study aims to provide insights into the most suitable intervention that can optimize the examination process, improve examination success rates, and minimize potential discomfort or distress experienced by infants.

It is anticipated that the results of this study will inform healthcare professionals and researchers about the benefits of auditory stimulation (white noise) and the additional advantages of multisensory stimulation during retinopathy examinations. Ultimately, this research aims to enhance the overall quality of care provided to premature infants, leading to improved visual outcomes and long-term well-being for this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Premature newborns with a gestational age of ≤ 32 weeks or newborns with a birth weight of < 1500 g, according to the records.
* Neonates undergoing a first-time eye exam to screen for retinopathy of prematurity.
* Newborns with their mother.
* Newborns who have not been fed in the last hour.

Exclusion Criteria:

* Newborns who need cardiopulmonary resuscitation (CPR) during the exam.
* Newborns experiencing apnea at the time of examination

Ages: 32 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Neonatal Pain | first 30 minutes during procedure
  The Premature Infant Pain Profile (PIPP) is a validated and widely used tool designed to assess pain in preterm infants. It takes into account physiological and behavioral indicators that are indicative of pain in this population. The PIPP scale includes the evaluation of facial expressions, gestational age, heart rate, oxygen saturation, and behavioral state to assess pain levels. Accordingly, the highest is 21 points and the lowest is 0 points. If the Premature Baby Pain Profile is between 0-6 points, the pain is considered mild, 7-12 points moderate, 13-21 points severe.

CONTACTS AND LOCATIONS:
Overall Officials: Halil İbrahim HI Taşdemir, PhD, Study Director — Burdur Mehmet Akif Ersoy University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
will be decided later